CLINICAL TRIAL: NCT06928740
Title: Evaluation de l'efficacité Sur l'anxiété de l'Application numérique Musicale, Music Care® Versus MEOPA, Kalinox® Chez Des Patients bénéficiant d'Une Infiltration Lombaire scanoguidée. Etude Monocentrique contrôlée randomisée de Non infériorité en Ouvert.
Brief Title: Efficacy on Anxiety of the Digital Music Application Versus Equimolar Mixture of Oxygen and Nitrous Oxide in Patients Receiving CT-guided Lumbar Infiltration
Acronym: MKI-TDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2024-2/FT01
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain; Anxiety
Keywords: Music therapy; Computerized tomography scan; ENOMO; Radiographer
MeSH Terms: conditions — Low Back Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Care (Experimental)
  Interventions: Other: Music Care® device
- Control (Active Comparator)
  Interventions: Other: EMONO

INTERVENTIONS:
Other: Music Care® device — Installation of the Music Care® device, selection of the sequence based on the patient's musical taste, listening to at least 20-minute sequence in the preparation room. Once placed on the scanner table, the patient listens to the same sequence as in the preparation room.
  Arms: Music Care
Other: EMONO — Equimolar mixture of oxygen and nitrous oxide given as usual care
  Arms: Control

SUMMARY:
Since the Covid-19 crisis, patients appear more stressed, with increasing fear of exams and the hospital environment, in particular for CT scan teams, which require injections. Currently, an equimolar mixture of oxygen and nitrous oxide (EMONO) is used to calm patients. However, the patient's prone position complicates its use, with patients sometimes in painful position and the discomfort of gas inhalation (nausea, dizziness, etc.), as well as reduced lung capacity. Greater patient anxiety increases the risk of complications, or even failure, (unexpected movement, stiffness, refusal to complete the procedure, etc.). In this study, music therapy using Music Care® tablets, was tested to replace EMONO. The study authors hypothesize that the use of the Music Care® device will have a comparable efficacy to that of EMONO (non-inferiority) in reducing patient anxiety during CT-guided lumbar infiltration. Furthermore, the study authors hypothesize that this simple, non-invasive method, with no contraindications for the patient, will be better tolerated and appreciated by both the patient and the paramedical team in charge of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with low back pain and an indication for CT-guided foraminal, posterior joint, or pudendal injection
* Patient with an anxiety score ≥ 35/100 based on the STAI-ETAT questionnaire

Exclusion Criteria:

* The subject is participating in another drug or category I interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient who has already received a CT-guided posterior articular, foraminal, epidural, or pudendal injection
* Indication for epidural or cervical injection
* Patient who is deaf or hard of hearing
* Contraindications to EMONO
* Facial or head trauma making it impossible to wear a nasofacial mask or headphones
* Patient who has taken an anxiolytic medication within 24 hours prior to the injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety between groups | Baseline
  0-100 visual analog scale (VSA)
Anxiety between groups | Day 0: upon locating helix and a skin location
  0-100 visual analog scale (VSA)
Anxiety between groups | Day 0: before injection of corticosteroids
  0-100 visual analog scale (VSA)

SECONDARY OUTCOMES:
Patient satisfaction between groups | Day 0: Before discharge from imagery department
  0-100 visual analog scale (VSA)
Patient comfort between groups | Day 0: After injection of corticosteroids
  0-100 visual analog scale (VSA)
Patient-reported pain between groups | Day 0: Before injection of corticosteroids
  0-100 visual analog scale (VSA)
Patient-reported pain between groups | Day 0: After injection of corticosteroids
  0-100 visual analog scale (VSA)
Anxiety between groups according to type of injection (foraminal, pudendal or posterior articular) | Day 0: Before injection of corticosteroids
  0-100 visual analog scale (VSA)
Anxiety between groups according to type of injection (foraminal, pudendal or posterior articular) | Day 0: After injection of corticosteroids
  0-100 visual analog scale (VSA)
Satisfaction of radiographer between groups | Day 0
  0-100 visual analog scale (VSA)
Rate of adverse events between groups | Day 0: During procedure
  According to Common Terminology Criteria for Adverse Events version 5.0 (grade 1-5)
Rate of adverse events between groups | Day 0: immediately after procedure
  According to Common Terminology Criteria for Adverse Events version 5.0 (grade 1-5)
Rate of complications between groups | Day 0: During procedure
  According to Clavien-Dindo (grade I-V)
Rate of complications between groups | Day 0: immediately after procedure
  According to Clavien-Dindo (grade I-V)

CONTACTS AND LOCATIONS:
Overall Officials: Florelle TERRA, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nimes, Nîmes, France